CLINICAL TRIAL: NCT02710331
Title: Ethanol and Cannabinoid Effects on Simulated Driving and Related Cognition: Substudy III
Acronym: THC-ETOH-III
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015208.C
Record Dates: First submitted 2016-03-10; First posted 2016-03-16 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cannabis; Alcohol Effect; Driving Under the Influence of Alcohol and Other Drugs
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active THC and Placebo Ethanol (Experimental)
  Interventions: Drug: Active Dronabinol; Drug: Placebo
- Active THC and Active Ethanol (Experimental)
  Interventions: Drug: Active Dronabinol; Drug: Active Ethanol
- Placebo THC and Active Ethanol (Experimental)
  Interventions: Drug: Placebo; Drug: Active Ethanol
- Placebo THC and Placebo Ethanol (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Dronabinol — 10 mg capsule of Dronabinol will be administered orally.
  Arms: Active THC and Active Ethanol; Active THC and Placebo Ethanol
Drug: Placebo — Control: no alcohol, administered for ~80 minutes.
  Arms: Active THC and Placebo Ethanol; Placebo THC and Placebo Ethanol
Drug: Placebo — Control: Placebo pill (no active cannabinoids) administered orally.
  Arms: Placebo THC and Active Ethanol; Placebo THC and Placebo Ethanol
Drug: Active Ethanol — Target BrAC of 0.04% reached over 20 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 2 drinks over 1 hour. Administered over a total of 80 minutes.
  Arms: Active THC and Active Ethanol; Placebo THC and Active Ethanol

SUMMARY:
The overarching goal of this study is to characterize the effects of ethanol and cannabinoids on simulated driving and related cognition.

DETAILED DESCRIPTION:
To study the effects of ethanol clamped at BAC 0.04% (equivalent to consuming approximately 2 drinks over 1 hour) and oral Dronabinol (10 mg capsule) on driving.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 21 to 55 years of age (extremes included).
* Exposed to cannabis at least once.
* Exposed to alcohol at least once.
* Able to provide informed consent.

Exclusion Criteria:

* Cannabis naïve
* Alcohol naïve
* Positive pregnancy screen
* Hearing deficits
* Sesame oil allergy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline: Road Tracking Error | baseline, +100, +210 mins after start of dronabinol administration

SECONDARY OUTCOMES:
Change from Baseline: Biphasic Alcohol Effects Scale (BAES) | baseline, +60, +90, +210, +360 mins after start of dronabinol administration
  A scale designed to assess the stimulant and sedative effects associated with alcohol intoxication.
Change from Baseline: Visual Analog Scale (VAS) | baseline, +60, +90, +210, +360 mins after start of dronabinol administration
  Feeling states associated with alcohol and cannabis intoxication will be measured using this self-report scale of feeling states.
Change from Baseline: Cognitive Test Battery | baseline, +120 mins after start of dronabinol administration
  Several computer tasks will be administered to assess alcohol and THC effects on driving related cognition, including:
  visual vigilance, visual motor function, attention and working memory, and processing speed.
Change from Baseline: Willingness to Drive Scale | baseline, +60, +90, +210, +360 mins after start of dronabinol administration
  Subjects will be asked to rate their willingness to drive at their current state in the context of various scenarios including willingness to drive from testing facility to a number of destinations that are different driving distances.
Change from Baseline: Number of Joints Scale | baseline, +60, +90, +210, +360 mins after start of dronabinol administration
  Subjects will be asked to rate the number of standard joints that they believe they have been administered.
Change from Baseline: Number of Drinks Scale | baseline, +60, +90, +210, +360 mins after start of dronabinol administration
  Subjects will be asked to rate the number of standard drinks that they believe they have been administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit, VA Connecticut Healthcare System, West Haven, Connecticut, United States